CLINICAL TRIAL: NCT05271344
Title: Standard Preoperative Oral Immunonutrition Versus Oral Immunonutrition With Synbiotics, Sustained Omega 3 Impregnation and Vitamin D in Patients Undergoing Duodenopancreatectomy for Tumoral Lesion : a Prospective, Placebo-controlled, Double-blind, Randomized Clinical Trial. The SIO3D Study.
Brief Title: Oral Immunonutrition With Synbiotics, Omega 3 and Vitamin D in Patients Undergoing Duodenopancreatectomy for Tumoral Lesion.
Acronym: SIO3D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, Alain Pans, Head of Clinic, Department of Abdominal Surgery and Transplantation, Centre Hospitalier Universitaire de Liege
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SIO3D
Record Dates: First submitted 2022-01-26; First posted 2022-03-09 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Pancreatic Cancer; Complication,Postoperative; Surgery
Keywords: synbiotics; omega 3; vitamin D; probiotics; prebiotics
MeSH Terms: conditions — Pancreatic Neoplasms; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Placebo products for probiotics, prebiotics, omega 3 and vitamin D
  Interventions: Dietary Supplement: Nutritional Products
- Treated Group (Experimental): Omega 3 fatty acids for 7 days (before starting conventional oral immunonutrition supplement), Probiotics for 14 days before and after the operation, Prebiotics for 14 days before and after the operation, Vitamin D for 6 days before the operation.
  Interventions: Dietary Supplement: Nutritional Products

INTERVENTIONS:
Dietary Supplement: Nutritional Products — Omega 3 : 1 softgel, 3 x/d Probiotics : 1 caps / d Prebiotics : 1 measuring spoon of powder to be diluted in water, 1x/d Vitamin D : 1 tablet, 2x/d

SUMMARY:
The purpose of this trial is to demonstrate that synbioimmunonutrition (SI) combined with omega-3 fatty acids (O3) and Vitamin D (D) is superior to conventional 7-day preoperative immunonutrition in terms of reducing overall morbidity, in cases of duodenopancreatectomy for tumoral lesion.

DETAILED DESCRIPTION:
To the best knowledge of the Investigators, a comprehensive multimodal approach to reduce postoperative morbidity in duodenopancreatectomies has not yet been evaluated. In the study, the Investigators combine the main nutritional interventions currently available and already having an individual scientific basis, sequentially and simultaneously, for a potential synergistic effect.

In cases of duodenopancreatectomy for tumoral lesion, a group of patients taking only conventional immunonutrition regimen (CIR), for 7 preoperative days, will be compared with a second group where immunonutrition will be maximised by the addition of omega 3 for 1 week prior to the administration of CIR, synbiotics for 14 days pre- and post-operatively, and preoperative vitamin D supplementation for 6 days, in terms of postoperative overall morbidity.

ELIGIBILITY:
Inclusion Criteria:

* All cases of duodenopancreatectomy for tumoral lesions.

Exclusion Criteria:

* Distal or total pancreatectomies, as well as procedures for chronic pancreatitis
* Patient refusal or inability to provide informed consent
* Use of dietary supplements containing omega 3, pre- or probiotics within 15 days prior to protocol initiation
* Severe cardiorespiratory or renal insufficiency
* HIV
* Cirrhosis Child-Pugh B-C
* Inability to feed by mouth
* Intestinal obstruction
* Unresectable tumor or metastatic disease on preoperative work-up
* Cardiac valvular pathology
* Short bowell syndrome
* Haemophilia
* Known allergy or intolerance to fish oil, fish or shellfish, milk, soy or components of the products used
* BMI < 16kg/m2
* Weight loss > 15% in the last 6 months
* Little or no food in the last 10 days
* Hypercalcemia
* Pregnancy, breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Calculation of the Comprehensive Complication Index (CCI) | From the Day of the operation to the patient's discharge Day of the hospital, up to 90 days after surgery
  This criterion takes into account all the complications of a given patient by weighting their relative importance. It varies from 0 to 100. A score of 0 means the absence of complications. A score of 100 is the death.

SECONDARY OUTCOMES:
Rate of infectious or non infectious complications and rate of mortality | up to 90 days after surgery
  Wound infection, pulmonary infection, urinary infection, intra-abdominal abscess, sepsis, pancreatic fistula, delayed gastric emptying, wound dehiscence, intestinal obstruction, intra-abdominal bleeding, pulmonary embolism, ...
Research of occult-bacterial translocation in blood samples | Day+1 and Day+4 postoperative day
  q-PCR technique
Metagenomic characterization of the faecal microbiota | Day-19 (or Day-18, or Day-17, or Day-16) preoperative day and Day-1 preoperative day
  Metagenomic sequencing through faecal samples
Blood determination of lipopolysaccharide binding protein | Day-19 (or Day-18, or Day-17, or Day-16) preoperative day and the day of the operation
  As a measure of intestinal barrier integrity

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud De Roover, Pr, Study Director — Centre Hospitalier Universitaire de Liege; Alain Pans, MD, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (1):
- CHU, Liège, Belgium

REFERENCES:
- [Background] Jablonska B, Mrowiec S. The Role of Immunonutrition in Patients Undergoing Pancreaticoduodenectomy. Nutrients. 2020 Aug 23;12(9):2547. doi: 10.3390/nu12092547. PMID 32842475